CLINICAL TRIAL: NCT01653015
Title: A Randomized Controlled Trial of Live Attenuated Vaccine Versus Trivalent Inactivated Vaccine in Hutterite Children
Brief Title: Live Versus Inactivated Influenza Vaccine Study in Hutterite Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RC1-274129
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine LAIV (Experimental): Live attenuated influenza vaccine (LAIV).
  Interventions: Biological: Trivalent Inactivated Vaccine
- Influenza vaccine TIV (Active Comparator): Trivalent inactivated vaccine (TIV).
  Interventions: Biological: Live Attenuated Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Vaccine — Influenza vaccination, 0.5 ml dose administered intramuscularly. Previously unvaccinated children who are less than 9 years of age at the time of immunization will receive a second 0.5 ml dose four weeks later.
  Other Names: VAXIGRIP by Sanofi Pasteur
  Arms: Influenza vaccine LAIV
Biological: Live Attenuated Influenza Vaccine — Influenza vaccination, 0.2 ml dose administered intranasally. Previously unvaccinated children who are less than 9 years of age at the time of immunization will receive a second 0.2 ml dose of the vaccine four weeks later.
  Other Names: FLUMIST by Mediummune.
  Arms: Influenza vaccine TIV

SUMMARY:
There is uncertainty about whether a live attenuated vaccine (LAIV) offers additional benefit over inactivated trivalent influenza vaccine (TIV) in providing indirect benefit to those who are unvaccinated through herd immunity. The goal of this randomized clinical trial is to determine whether immunizing children in Hutterite colonies with LAIV can provide increased community-wide protection over TIV. Children aged 3 to 15 years in Hutterite colonies from Alberta and Saskatchewan will be randomized to one of two regimens: TIV or LAIV. The primary outcome of this study will be laboratory-confirmed influenza as detected by PCR in all participants (i.e vaccine recipients and nonrecipients). Secondary outcomes will include influenza-like illness, hospitalization, pneumonia, death, antibiotic use, absenteeism.

DETAILED DESCRIPTION:
The goal of this study is to test whether immunizing children in Hutterite colonies with LAIV can significantly reduce laboratory-confirmed influenza in the entire community compared to TIV. We hypothesize that ≥70% uptake of LAIV compared to a similar uptake of TIV among healthy children and adolescents will reduce laboratory-confirmed influenza in LAIV colonies by 50% compared to TIV colonies. Other specific objectives are to determine if LAIV reduces influenza in the healthy children and adolescents immunized and if LAIV reduces the following relative to TIV in all participants: influenza-like illness, antimicrobial prescriptions, physician-diagnosed otitis media, school or work-related absenteeism, physician visits for respiratory illness, lower respiratory infection, pneumonia, hospitalizations, and death. We will assess reactogenicity in both study groups.

ELIGIBILITY:
Group A:

Inclusion criteria:

* healthy children and adolescents aged 36 months to 15 years who will be immunized as part of the intervention.

Exclusion criteria:

1. anaphylactic reaction to a previous dose of LAIV or TIV
2. known IgE-mediated hypersensitivity to eggs manifested as hives, swelling of the mouth and throat, difficulty in breathing, hypotension, or shock
3. history of asthma
4. medically diagnosed or treated wheezing within 42 days before enrollment
5. Guillain-Barré syndrome within eight weeks of a previous influenza vaccine
6. anaphylactic reaction to gentamicin
7. anaphylactic reaction to gelatin
8. anaphylactic reaction to neomycin
9. anaphylactic reaction to arginine
10. pregnancy
11. household contact who is severely immunocompromised being cared for in a protective environment (i.e hematopoietic stem cell transplant)
12. use of aspirin or salicylate-containing products within 30 days before enrollment.

Group B:

Inclusion Criteria

* other Hutterite community members that are not in Group A

Exclusion Criteria:

* there are no exclusion criteria for this category of participants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4611 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza infection. | up to 3 years

SECONDARY OUTCOMES:
Influenza like illness. | December to June each year for 3 years.
Physician diagnosed otitis media. | December to June each year for 3 years.
Antimicrobial prescriptions. | December to June each year for 3 years.
School or work related absenteeism. | December to June each year for 3 years.
Physician visits for respiratory illness. | December to June each year for 3 years.
Lower respiratory infection or pneumonia. | December to June each year for 3 years.
Hospitalization for lower respiratory infection or pneumonia. | December to June each year for 3 years.
All cause hospitalizations. | December to June each year for 3 years.
Deaths due to lower respiratory infections or pneumonia. | December to June each year for 3 years.
All cause deaths. | December to June each year for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Loeb M, Russell ML, Manning V, Fonseca K, Earn DJ, Horsman G, Chokani K, Vooght M, Babiuk L, Schwartz L, Neupane B, Singh P, Walter SD, Pullenayegum E. Live Attenuated Versus Inactivated Influenza Vaccine in Hutterite Children: A Cluster Randomized Blinded Trial. Ann Intern Med. 2016 Nov 1;165(9):617-624. doi: 10.7326/M16-0513. Epub 2016 Aug 16. PMID 27538259